CLINICAL TRIAL: NCT06723496
Title: Psychiatric Problems in Children With Acute Lymphoblastic Leukemia and Their Caregivers in South Egypt Cancer Institute
Brief Title: Psychiatric Problems in Children With Acute Lymphoblastic Leukemia and Their Caregivers
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer of neurology and psychiatry department, Assiut University
Other Study IDs: psych-oncology
Record Dates: First submitted 2024-11-29; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia ALL
Keywords: psychiatry; children; caregivers; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: children with ALL
  Interventions: Behavioral: Child Behavioral Checklist (CBCL):is a checklist parents complete to detect emotional and behavioral problems in children and adolescent, it consists of 113 questions for both groups.; Behavioral: parent report on child's responses to stress (PCT):is a questionnaire which is used to obtain mothers' and fathers' reports of their children's coping with cancer; Behavioral: Symptom Checklist -90- Revised (SCL-90-R) for parents; Behavioral: posttraumatic stress disorders by posttraumatic check list -5 (PCL-5) for parents
- healthy control group
  Interventions: Behavioral: Child Behavioral Checklist (CBCL):is a checklist parents complete to detect emotional and behavioral problems in children and adolescent, it consists of 113 questions for both groups.; Behavioral: Symptom Checklist -90- Revised (SCL-90-R) for parents

INTERVENTIONS:
Behavioral: Child Behavioral Checklist (CBCL):is a checklist parents complete to detect emotional and behavioral problems in children and adolescent, it consists of 113 questions for both groups. — is a checklist parents complete to detect emotional and behavioral problems in children and adolescent, it consists of 113 questions.
Behavioral: parent report on child's responses to stress (PCT):is a questionnaire which is used to obtain mothers' and fathers' reports of their children's coping with cancer — It includes a list of 12 cancer -related stressors (e.g., missing school, frequent hospital or clinic visits, changes in personal appearance), and 57 items reflecting voluntary (coping) and involuntary (automatic) stress responses of children /adolescents in response to cancer-related stressors
  Groups: cases group
Behavioral: Symptom Checklist -90- Revised (SCL-90-R) for parents — It is a method to evaluate psychological problems and identify symptoms, it includes 90 symptoms and evaluate nine symptomatic dimensions
Behavioral: posttraumatic stress disorders by posttraumatic check list -5 (PCL-5) for parents — It is a 20 -item measure that assess the 20 DSM-5 symptoms of PTSD.
  Groups: cases group

SUMMARY:
Cancer in childhood represents a significant health challenge, with approximately 400,000 children and adolescents aged 0-19 years diagnosed annually. The oncological landscape of pediatric populations is characterized by diverse malignancies, with leukemias, brain cancers, lymphomas, and solid tumors such as neuroblastoma and Wilms tumors constituting the predominant diagnostic categories. Among these, acute lymphoblastic leukemia (ALL) emerges as the most prevalent childhood malignancy.

Historically, a cancer diagnosis portended an almost invariably fatal outcome. However, contemporary medical interventions have dramatically transformed this narrative. Since 1980, mortality rates across pediatric cancer types have declined by more than 50%, representing a remarkable advancement in clinical oncology. Notably, ALL demonstrates an exceptionally optimistic prognosis, with over 90% of patients achieving complete remission.

Despite these encouraging survival statistics, the cancer experience extends beyond physiological parameters. Children diagnosed with leukemia and their familial support systems frequently encounter complex psychological challenges. These manifestations encompass a spectrum of emotional responses, including anxiety, shock, denial, depression, and adaptive difficulties. Critically, these psychological sequelae are not confined to the diagnostic and treatment phases but often persist even after disease remission

The multidimensional nature of the cancer experience prompted the emergence of a specialized subdiscipline in 1992. Termed "psycho-oncology" in the United States and "psychosocial oncology" predominantly in European contexts, this field addresses two fundamental psychological dimensions:

Emotional and psychosocial responses of patients, families, and caregivers throughout the disease trajectory Psychological, behavioral, and social factors potentially influencing cancer morbidity and mortality.

Consequently, contemporary pediatric oncological care adopts a holistic paradigm. The therapeutic objective transcends mere physical restoration, aspiring to ensure the comprehensive social and emotional well-being of both the child and the familial ecosystem.

ELIGIBILITY:
A) Case groups:

1. The patients:

Inclusion criteria: the investigators included children with the following criteria:

* Newly diagnosed with ALL
* Aged 6 to 18 years old.

Exclusion criteria: the investigators excluded children with following criteria:

• Children with malignancies other than ALL.

* Age <6 years old and >18 years old.
* Children with chronic illness e.g., diabetes mellitus, inflammatory bowel disease, congenital heart disease, cerebral palsy, etc.
* Children with history of psychiatric illness or intellectual disability.

  2 -the caregivers:

Inclusion criteria:

* The caregivers who are in charge of the case children during treatment.

Exclusion criteria:

• The caregivers with history of psychiatric illness.

B) Control groups:

1. the control children:

   Inclusion criteria:

   • Children with matched age and gender to case group.

   Exclusion criteria:
   * Children with history of having malignancy or current malignancy.
   * Children with history of medical, chronic illness or psychiatric disorders.
2. the control caregivers:

Inclusion criteria:

• Caregivers with matched age and gender to the caregivers' case group.

Exclusion criteria:

• Caregivers with history of psychiatric illness.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators will recruit two groups; first group will be new cases with ALL with their caregivers attending outpatient clinic or admitted inpatient oncological ward and the second group will be healthy control children with their caregivers.
  Regarding cases group, every patient will be followed for 6 months with the assessment at diagnosis, post induction phase, post consolidation phase and after 3months from the beginning of the maintenance phase.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of psychiatric comorbidity in children with ALL and their caregivers at different stages of illness at South Egypt cancer institute | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Assiut university,Assiut,Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spinetta JJ, Jankovic M, Masera G, Ablin AR, Barr RD, Ben Arush MW, D'Angio GJ, Van Dongen-Melman J, Eden T, Epelman C, Martins AG, Greenberg ML, Kosmidis HV, Oppenheim D, Zeltzer PM. Optimal care for the child with cancer: A summary statement from the SIOP Working Committee on Psychosocial Issues in Pediatric Oncology. Pediatr Blood Cancer. 2009 Jul;52(7):904-7. doi: 10.1002/pbc.21863. PMID 19142992
- [Background] Holland JC. Psycho-oncology: Overview, obstacles and opportunities. Psychooncology. 2018 May;27(5):1364-1376. doi: 10.1002/pon.4692. PMID 29749682